CLINICAL TRIAL: NCT00655395
Title: A Phase I/Phase II Evaluation of Laromustine (VNP40101M), A Sulfonylhydrazine Alkylating Agent, Combined With Infusional Cytarabine in Elderly Patients With Acute Myeloid Leukemia and High Risk Myelodysplastic Syndrome
Brief Title: Treatment of Elderly Patients With Acute Myeloid Leukemia (AML) and High Risk Myelodysplastic (MD) Syndrome With Laromustine and Infusional Cytarabine
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Viron Therapeutics Inc (Industry)
Collaborators: Vion Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0702009008; VNP40101M
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2018-08

CONDITIONS: Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome (MDS)
Keywords: Leukemia; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia | interventions — laromustine; Cytarabine

ARMS (5):
- 1 (Experimental): 1. Laromustine 300 mg/m2 (cohort 1) IV on day 1 over 30 - 60 minutes. Laromustine will be administered approximately 3-4 hours following the start of infusional Ara C.
  2. Ara C at 100 mg/m2/day as a continuous infusion daily for 7 days. Appropriate antiemetics are given during the Ara C infusion.
  Interventions: Drug: Laromustine (VNP40101M) and Ara-C
- 2 (Experimental): 1. Laromustine 400 mg/m2 (cohort 2) IV on day 1 over 30 - 60 minutes. Laromustine will be administered approximately 3-4 hours following the start of infusional Ara C.
  2. Ara C at 100 mg/m2/day as a continuous infusion daily for 7 days. Appropriate antiemetics are given during the Ara C infusion.
  Interventions: Drug: Laromustine (VNP40101M) and Ara-C
- 3 (Experimental): 1. Laromustine 500 mg/m2 (cohort 3) IV on day 1 over 30 - 60 minutes. Laromustine will be administered approximately 3-4 hours following the start of infusional Ara C.
  2. Ara C at 100 mg/m2/day as a continuous infusion daily for 7 days. Appropriate antiemetics are given during the Ara C infusion.
  Interventions: Drug: Laromustine (VNP40101M) and Ara-C
- 5 (Experimental): 1. Laromustine will be administered at the recommended phase II dose on day 1 over 30 - 60 minutes. Laromustine will be administered approximately 3-4 hours following the start of infusional Ara C.
  2. Ara C at 100 mg/m2/day as a continuous infusion daily for 7 days. Appropriate antiemetics are given during the Ara C infusion.
  Interventions: Drug: Laromustine (VNP40101M) and Ara-C
- 4 (Experimental): 1. Laromustine 600 mg/m2 (cohort 4) IV on day 1 over 30 - 60 minutes. Laromustine will be administered approximately 3-4 hours following the start of infusional Ara C.
  2. Ara C at 100 mg/m2/day as a continuous infusion daily for 7 days. Appropriate antiemetics are given during the Ara C infusion.
  Interventions: Drug: Laromustine (VNP40101M) and Ara-C

INTERVENTIONS:
Drug: Laromustine (VNP40101M) and Ara-C — 1. Laromustine 300 mg/m2 (cohort 1), 400 mg/m2 (cohort 2), 500 mg/m2 (cohort 3) IV on day 1 over 30 - 60 minutes. Laromustine will be administered approximately 3-4 hours following the start of infusional Ara C.
  2. Ara C at 100 mg/m2/day as a continuous infusion daily for 7 days. Appropriate antiemetics are given during the Ara C infusion.

SUMMARY:
* The purpose of the Phase I portion of this study is to evaluate the safety of this combination of medications and to determine the appropriate dose of VNP40101M to be used in combination with infusional cytarabine (araC) in elderly patients with Acute Myeloid Leukemia (AML) and High Risk Myelodysplastic Syndrome (MDS).
* The purpose of the Phase II portion of the study is to evaluate the effectiveness (overall response rate) for patients treated with VNP40101M and infusional cytarabine induction therapy.

DETAILED DESCRIPTION:
There is no known standard chemotherapy that is considered effective for older patients with AML or high risk MDS at this time, and with current treatment, tumor reduction can be difficult to achieve and is short-lived. We are, therefore, interested in developing new drugs that might have a longer-lasting effect against disease.

Laromustine is a new drug that has been shown to have anti-cancer activity in animal and human studies. It interacts with the DNA of a cancer cell and kills the cell. Cytarabine (AraC) is a commercially available chemotherapy drug that is active against leukemia and used routinely when the disease is first diagnosed. In previous studies, when higher doses of laromustine were given, laromustine and AraC achieved more responses than patients treated with AraC alone. However, this advantage was offset by the fact that more patients given laromustine/AraC died to due side effects. We wish to determine the effectiveness of laromustine in combination with infusional AraC in AML and high risk MDS patients who are 60 or more years of age.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML based on WHO criteria (greater than 20% blasts in the bone marrow or blood) excluding AML M3, acute promyelocytic leukemia OR diagnosis of high-risk MDS defined as International Prognostic Scoring System INT-2.
* ECOG performance status equal to 0, 1, 2.
* No prior treatment for AML with myeloablative treatment. Patients may have prior treatment with a biologic therapy. Patients with MDS or AML that has evolved from MDS could have received prior low-dose cytotoxic therapy with agents such as azacytidine or low-dose Ara C.
* Ability to sign an Informed Consent according to institutional guidelines.
* Patients must have the following clinical laboratory values within 24 hours prior to beginning protocol treatment: a) serum creatinine less than or equal to 2.0mg/dl. b) total bilirubin less than or equal to 2.0 mg/dl c) ALT or AST less than or equal to 5 times the upper limit of normal.

Exclusion Criteria:

* Uncontrolled active infection. Patients with infections who are under active treatment with antibiotics and whose infections are controlled may be entered into the study. Patients with chronic hepatitis are eligible.
* Active heart disease including myocardial infarction, symptomatic coronary artery disease, arrhythmias not controlled by medication or uncontrolled congestive heart failure.
* Severe pulmonary disease not controlled with medication.
* Patients with serum creatinine > 2.0, serum bilirubin > 2.0. ALT or AST greater that 5 times the upper limit of normal. Patients with bilirubin or creatinine outside the acceptable levels will be considered eligible if this abnormality is clearly leukemia related and discussed with the principal's investigator prior to enrollment.
* Patients concurrently receiving any other standard or investigational treatment for leukemia with the exception of hydroxyurea.
* Since the formulation contains 30% ethanol, patients being treated with Antabuse (disulfiram) are excluded from the study.
* Patients with APL t(15;17)
* Patients with ECOG performance status of 3 or 4.
* Patients should be off metronidazole (Flagyl) at least 24 hours before starting laromustine.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2010-04 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The objectives of this study are to evaluate the safety and efficacy of VNP40101M in combination with infusional Ara C as induction therapy in elderly patients with AML or high-risk MDS evolving to AML. | Subjects will be closely monitored continuously throughout the study.

SECONDARY OUTCOMES:
The secondary objective of this study is to evaluate this regimen for toxicities in this elderly population. | Subjects will be closely monitored continuously throughout the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Weill Cornell Medical College, New York, New York, United States